CLINICAL TRIAL: NCT01337921
Title: A Randomized Controlled Trial on a Multi-strain Synbiotic vs. a Multi-strain Probiotic on Fecal Colonization in the Very Low Birth Weight Infant
Brief Title: A Multi-strain Synbiotic Versus a Multi-strain Probiotic in Premature Infants
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Pending further safety information regarding polysaccharides and premature infants
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 0065-11-FB
Record Dates: First submitted 2011-03-16; First posted 2011-04-19 (Estimated); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Feeding; Difficult, Newborn; Necrotizing Enterocolitis
MeSH Terms: conditions — Enterocolitis, Necrotizing | interventions — Lacteol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Multi-strain Synbiotic (Experimental): Multi-strain probiotic with prebiotics
  Interventions: Dietary Supplement: Multi-strain Probiotic
- Multi-strain Probiotic (Active Comparator): Multi-strain Probiotic without prebiotics.
  Interventions: Dietary Supplement: Multi-strain Probiotic

INTERVENTIONS:
Dietary Supplement: Multi-strain Probiotic — Multi-strain Synbiotic: 1.5 billion CFU of Lactobacillus acidophilus, Bifidobacterium bifidum,and Bifidobacterium lactis WITH galacto-oligosaccharide(GOS)/fructo-oligosaccharide (FOS) combination at 1g/dL (0.9g/dL GOS/ 0.1g/dL FOS)
  Other Names: Lactobacillus

SUMMARY:
The aims are to 1) compare two probiotic treatments (multi-strain synbiotic vs. multi-strain probiotic) on bifidobacteria fecal colonization counts at 1, 2, 3, and 4 weeks of life, 34 weeks corrected gestation age (CGA) ; 2) compare infants successfully colonized with probiotic organisms to infants not successfully colonized at 1, 2, 3, and 4 weeks of life, 34 weeks CGA on infant outcomes and on stress biomarker patterns at birth, day of life (DOL) 1, DOL 7; 3) determine long-term safety and outcomes of probiotic treatments at 6, 16, and 24 months CGA.

DETAILED DESCRIPTION:
Feeding Intolerance and other GI issues are a major concern in a NICU hospitalized population. Successful colonization with probiotic bacteria is thought to impact the incidence of GI related issues. This study will study the impact of prebiotics on the colonization of a population of VLBW infants in the NICU setting.

ELIGIBILITY:
Inclusion Criteria:

* infants with a birth weight < 1500g
* admission to NICU at The Nebraska Medical Center

Exclusion Criteria:

* infants who have congenital anomalies
* have a diagnosis of a congenital metabolic disease
* are made a ward of the State or
* are born to a mother < 19 years of age

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-06 (Estimated); Primary Completion 2011-06-16 (Actual); Study Completion 2011-06-16 (Actual)

PRIMARY OUTCOMES:
Comparing a multi-strain synbiotic vs. a multi-strain probiotic on mean bifidobacteria fecal colonization counts | 1,2, 3, 4 and 34 weeks of age
  Infants will be given the synbiotic or probiotic supplementation within the first week of life (upon inititation of enteral feedings) until approximately 34 weeks corrected gestational age.

SECONDARY OUTCOMES:
Compare the difference between two groups (multi-strain synbiotic vs. multi-strain probiotic) on demographic data and selected standard clinical infant outcomes. | From birth to NICU discharge (average 36 weeks corrected gestational age)
  Two probiotic groups will be compared on demographics: mean [birth wt(g), birth length(cm), birth hc(cm), GA at birth, 1-& 5- minute APGAR scores], race, gender, prenatal antibiotics(y/n), and enteral feeding type(breastmilk, formula, both); and on selected infant outcomes: Feeding Intolernce(number of times the feeding care plan is disrupted), NEC(y/n), late-onset sepsis(y/n), IVH(y/n;Grade I-IV), PDA(y/n), CLD(y/n), mean [endotracheal ventilation(days), inspired oxygen, discharge wt(g),discharge length(cm), discharge hc(cm), days to reach full feedings, length of stay, days on antibiotics].
Compare the difference between infants successfully colonized with probiotic organisms (>10^2 colonies on a 10^4-fold dilution plate)to infants not successfully colonized on demographics and selected standard clinical outcomes | 1 week of life to NICU discharge
  Two colonization groups will be compared on demographics: mean[birth wt(g), birth length(cm),birth hc(cm),GA at birth,1-& 5- minute APGAR scores],race, gender,prenatal antibiotics(y/n),and enteral feeding type(breastmilk, formula, both); and on selected infant outcomes: Feeding Intolernce(number of times the feeding care plan is disrupted), NEC(y/n), late-onset sepsis(y/n), IVH(y/n;Grade I-IV), PDA(y/n), CLD(y/n), mean [endotracheal ventilation(days), inspired oxygen, discharge wt(g),discharge length(cm), discharge hc(cm), days to reach full feedings, length of stay, days on antibiotics].
Compare infants successfully colonized with probiotic organisms(>10^2 colonies on a 10^4-fold dilution plate) to infants not successfully colonized on stress biomarker levels | day of life 1 to day of life 7
  Interquartile ranges of biomarkers will be compared between the two colonization groups. Biomarkers include: serum cortisol(cord blood), salivary cortisol (DOL 1,7), serum 8-hydroxydeoxyguanosine (cord blood), urinary 8-hydroxydeoxyguanosine (DOL 1,7)
Compare trends of stress biomarker levels in relation to demographics and selected standard infant outcomes | day of life 1 to day of life 7
  Interquartile ranges of biomarkers (listed above) will be compared on the demographic data and selected standard infant outcomes (listed above) at each time (DOL 1, 7) and over-time.
Compare the difference between the two probiotic treatment groups (multi-strain synbiotic vs. multi-strain probiotic) on longitudinal neurodevelopmental outcomes. | 6, 16 & 24 months corrected gestational age.
  Appropriate Bayley scales conducted by developmental pediatricians will be used for the neurodevelopmental data.

CONTACTS AND LOCATIONS:
Overall Officials: Ann Anderson-Berry, MD, Study Chair — University of Nebraska; Corrine K Hanson, PhD, Study Chair — UNMC